CLINICAL TRIAL: NCT05888233
Title: Allopurinol Improves Diastolic Function in African Americans With Resistant Hypertension
Brief Title: Allopurinol Improves Heart Function in African Americans With Resistant Hypertension
Acronym: RESIST
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F4655-P; I21RX004655-01 (NIH)
Record Dates: First submitted 2023-05-02; First posted 2023-06-05 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure Preserved Ejection Fraction; Resistant Hypertension
Keywords: Hypertension; Xanthine Oxidase; African American; Black; Heart Failure
MeSH Terms: conditions — Heart Failure, Diastolic; Hypertension; Heart Failure | interventions — Allopurinol

STUDY DESIGN:
Intervention Model Description: This is an open label unblinded drug pilot study to determine whether Allopurinol improves left ventricular diastolic function, exercise capacity, and quality of life in African American Veterans with resistant hypertension after 8-weeks of treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Allopurinol - African American Veterans (Experimental): Subjects will receive Allopurinol (300mg/daily) for 4 weeks. If tolerated, dose may be increased to 600mg/daily for an additional 4 weeks. Subjects will take Allopurinol (300-600mg/daily) for 8 weeks total
  Interventions: Drug: Allopurinol

INTERVENTIONS:
Drug: Allopurinol — Single arm of Allopurinol treatment for 300mg/daily for 4 weeks then may be increased to 600mg/daily for an additional 4 weeks.

SUMMARY:
African American adults in the United States have the highest prevalence rate of high blood pressure (hypertension) and heart failure in the world. African Americans with treatment resistant hypertension have higher levels of the enzyme - xanthine oxidase compared to Caucasians. This trial will test if administration of the xanthine oxidase inhibitor - Allopurinol (commonly used in the treatment of gout), given over a period of 8 weeks, will improve heart function, exercise ability and quality of life in African American Veterans with resistant hypertension.

DETAILED DESCRIPTION:
Hypertension among African American adults in the United States has one of the highest prevalence rates in the world and is related to adverse changes in left ventricular (LV) structure and function. Hypertension is an underlying factor in greater than 50% of African American adults with heart failure and is the strongest risk factor in that population. African American adults have a 50% increased incidence of heart failure, due in large part due to the greater prevalence and severity of hypertension.

Heart failure occurs 8 years earlier in African American adults compared with Caucasians. Further, African American adults with heart failure have worse quality of life and depressive symptoms and have a 5-year mortality rate that is 34% higher than in Caucasians. Although African American adults have the highest death rate for heart failure, they are consistently under-represented in clinical trials. The greater heart failure burden among African Americans calls for further work to discover effective preventive and therapeutic strategies for this higher-risk population with heart failure preserved ejection fraction (HFpEF).

An estimated 10-20% of hypertensive patients have resistant hypertension (RHTN), defined as having controlled or uncontrolled blood pressure with the use of 3 or more medications that includes a diuretic. A recent study reported increased plasma xanthine oxidase (XO) activity and mitochondrial DNA damage associated molecular products (mtDAMPs) levels in African American adults with RHTN, compared with Caucasian adults with RHTN. This supports the consensus that oxidative stress is higher in African American adults. Increased xanthine oxidase in heart muscle cells causes a breakdown of muscle structure and a decrease in calcium sensitivity, resulting in left ventricular (LV) dysfunction. A recent study shows that diastolic blood pressure, and other indices of LV diastolic function positively relate to xanthine oxidase activity among African American but not Caucasian RHTN patients.

Given the higher level of xanthine oxidase activity and mtDAMPs in African Americans, the purpose of this clinical trial is to test whether blockade with Allopurinol (for 8 weeks) will improve LV diastolic function, exercise capacity and quality of life metrics in 50 African American Veterans with resistant hypertension.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Veteran
2. African American
3. Resistant hypertension diagnosis (defined as blood pressure greater than 140/90 mmHg at 2 clinic visits despite the use of 3 antihypertensive medications at pharmacologically effective doses)
4. Locale - Birmingham, AL and surrounding areas

Exclusion Criteria:

1. History of heart failure
2. Chronic kidney disease (estimated creatinine clearance < 60 ml/min)
3. Chronic steroid therapy
4. Known coronary artery disease
5. Known causes of secondary hypertension
6. Already taking Allopurinol

Magnetic Resonance Imaging Exclusion

1. Claustrophobia
2. Cardiac implantable electronic device (permanent pacemaker and/or intracardiac defibrillator)
3. Metal clips and/devices or other item that specifically prohibit safe CMR

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Normalized peak early diastolic filling rate (E) | 8 weeks
  Change from baseline in left ventricular diastolic function index: Normalized peak early diastolic filling rate (E) after 8-weeks of treatment with Allopurinol. (Range 1.5 - 3.0 EDV/sec)
Six minute walk test | 8 weeks
  Change in exercise capacity by six minute walk test after 8-weeks of Allopurinol. Timed activity for distance walked (Distance range approximately 400-800m; Further distance = better outcome)
Self Reported health survey for Heart Failure | 8 weeks
  Change in self reported quality of life measures using Kansas City Heart Failure Questionnaire (KCCQ-12) after 8-weeks of Allopurinol. Scale (Minimum - 0 ; Maximum - 100; High score = worse outcome)
Self reported Health Survey | 8 weeks
  Change in self reported quality of life measures using the Quality of Life Medical Outcomes Study Questionnaire (SF 36 QOL) after 8-weeks of Allopurinol. Scale (Minimum - 0; Maximum - 100; High score = worse outcome)
Left ventricular end-diastolic volume index | 8 weeks
  Change from baseline in left ventricular diastolic function index: left ventricular end diastolic volume normalized to body surface area after 8-weeks of treatment with Allopurinol. (Range 40 - 100 mL/m2)
LV end-diastolic mass index | 8 weeks
  Change from baseline in left ventricular diastolic function index: LV end-diastolic mass indexed to body surface area after 8-weeks of treatment with Allopurinol. (Range: 40-100 grams/m2)
LV end-diastolic fractional shortening | 8 weeks
  Change from baseline in left ventricular diastolic function index: LV end-diastolic fractional shortening after 8-weeks of treatment with Allopurinol. (Range: 15-80%)
LV end-diastolic mid-wall radius to wall thickness ratio | 8 weeks
  Change from baseline in left ventricular diastolic function index: LV end-diastolic mid-wall radius to wall thickness ratio. Ratio (no units; Range: 1.5-4.0).
Normalized peak late diastolic filling rate (A), EDV/s | 8 weeks
  Change from baseline in left ventricular diastolic function index: Normalized peak late diastolic filling rate (A) after 8-weeks of treatment with Allopurinol. (Range 1.3 - 4.5 EDV/sec)

SECONDARY OUTCOMES:
Systolic Blood Pressure | 8 weeks
  Change in systolic blood pressure after 8 weeks of Allopurinol. Range: 120-200 mmHg
Xanthine Oxidase | 8 weeks
  Change in systemic levels of xanthine oxidase (range - Xanthine oxidase activity, U/mg protein - Range 0 - 0.1)
mitochondrial DNA damage-associated molecular patterns | 8 weeks
  Change in systemic levels of mitochondrial DNA damage-associated molecular patterns (range 0-5000 copies/uL)
Brain Natriuretic Peptide | 8 weeks
  Change in systemic levels of brain natriuretic peptide (BNP) after 8 weeks of Allopurinol (Scale 0 to > 100 pgmL; Minimum 0; Maximum >100).
Diastolic Blood Pressure | 8 weeks
  Change in diastolic blood pressure after 8 weeks of Allopurinol. Range: 70-110 mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Louis J Dellitalia, MD, Principal Investigator — Birmingham VA Medical Center, Birmingham, AL
Locations (1):
- Birmingham VA Medical Center, Birmingham, AL, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No